CLINICAL TRIAL: NCT01601925
Title: Distances From Cricoid Cartilage to the Targets of Stellate Ganglion Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, jong bum Choi, Yonsei University College of Medicine, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-2011-0231
Record Dates: First submitted 2012-05-03; First posted 2012-05-18 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Herpes Zoster; CRPS
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- neck extended group (Experimental): We measured the distances from cricoid cartilage to C6 or C7 transverse process in supine neutral and extended position of the neck.
  Interventions: Other: supine extended position of the neck

INTERVENTIONS:
Other: supine extended position of the neck — we measure the distances from cricoid cartilage to C6 or C7 transverse process in supine neutral and extended position of the neck

SUMMARY:
Stellate ganglion block targets are C6 transverse process or C7 transverse process in anterior paratracheal approach which is most popular method. Cricoid cartilage is known that it is located at C6 level in supine neutral position of the neck. But stellate ganglion block is performed in supine extended position of the neck. So cricoid cartilage will move up to cephalad direction and pain doctors should find C6 or C7 transverse process at lower neck area than cricoid cartilage.

ELIGIBILITY:
Inclusion Criteria:

* adults above age of 20 reserved for musculoskeletal ultrasonography

Exclusion Criteria:

1. past history of neck surgery
2. the limitation of neck motion due to rheumatoid arthritis, et al.
3. severe neck pain
4. inability to communicate or read or write

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-06 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
the distances from cricoid cartilage to C6, C7 transverse process in supine neutral and extended position of the neck | up to 1 week
  The distances from cricoid cartilage to C6, C7 transverse process will be measured in supine neural position and extended position of the neck up to 1 week after agreement to enroll

SECONDARY OUTCOMES:
the sexual difference in the distances from cricoid cartilage to C6, C7 transverse process in supine neutral or extended position of the neck | up to 1 week
  The sexual difference in the distances from cricoid cartilage to C6,C7 transverse process will be measured in supine neural position and extended position of the neck up to 1 week after agreement to enroll

CONTACTS AND LOCATIONS:
Overall Officials: Jong B Choi, Study Director — Yonsei University
Locations (1):
- Gangnam Severance hospital, Seoul, South Korea